CLINICAL TRIAL: NCT04437784
Title: Laparoscopic Versus Open Mesh Repair of Bilateral Primary Inguinal Hernia; 3 Armed Randomized Study
Brief Title: Laparoscopic Versus Open Mesh Repair of Bilateral Primary Inguinal Hernia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed El Messiry, Assistant professor of Surgery, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 302765
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Bilateral Inguinal Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sealed opaque envelopes containing computer generated random numbers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laparoscopic Trans-Abdominal Pre-Peritoneal (Lap TAPP group)) (Active Comparator): Both hernias were treated by laparoscopic trans-abdominal pre-peritoneal repair using 2 separate meshes fixed by endoscopic tackers
  Interventions: Procedure: Laparoscopic Trans-Abdominal Pre-Peritoneal
- Open Pre-Peritoneal Repair ( Open PP group) (Active Comparator): Both hernias were treated by open pre-peritoneal single mesh repair with suture fixation
  Interventions: Procedure: Open pre-peritoneal repair
- Bilateral Lichtenstein repair (LICHT group) (Active Comparator): treated by bilateral standard Lichtenstein repair using 2 separate meshes with suture fixation
  Interventions: Procedure: Bilateral Lichtenstein repair

INTERVENTIONS:
Procedure: Laparoscopic Trans-Abdominal Pre-Peritoneal — Laparoscopic trans-abdominal pre-peritoneal repair using 2 separate meshes fixed by endoscopic tackers
  Arms: Laparoscopic Trans-Abdominal Pre-Peritoneal (Lap TAPP group))
Procedure: Open pre-peritoneal repair — Open pre-peritoneal single mesh repair with suture fixation
  Arms: Open Pre-Peritoneal Repair ( Open PP group)
Procedure: Bilateral Lichtenstein repair — Bilateral standard Lichtenstein repair using 2 separate meshes with suture fixation
  Arms: Bilateral Lichtenstein repair (LICHT group)

SUMMARY:
The best approach for simultaneous repair of bilateral inguinal hernia is controversial. The aim of this study is to compare the outcomes after laparoscopic versus open mesh repair of bilateral primary inguinal hernia

DETAILED DESCRIPTION:
This prospective study included 180 patients with bilateral primary inguinal hernia; randomized by sealed envelopes into 3 groups; each includes 60 patients. Group I treated by laparoscopic trans-abdominal pre-peritoneal (TAPP) repair using 2 separate meshes, Group II treated by open pre-peritoneal (PP) single mesh repair, while Group III treated by bilateral Lichtenstein repair. The 3 groups were compared regarding: operative time, postoperative complications, postoperative pain, 3 years-recurrence rate and patient's satisfaction.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients with painless uncomplicated primary bilateral inguinal hernias

Exclusion Criteria:

* Immune compromised patients
* Coagulopathy
* Chronic liver or renal disease
* High-risk patients unfit for major surgery (ASA III or IV),
* Massive scrotal hernias, Recurrent or Complicated hernias
* Groin pain due to any other pathology
* Previous infra-umbilical surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Operative time | From skin incision until incision closure at the end of surgery
  Operative time (in minutes)
Postoperative pain after 24 hours | 24 hours after surgery
  Pain intensity was assessed 24 hours after surgery using the pain visual analogue scale (VAS) with values ranging from 1 (no pain) to 10 (worst possible pain)
Postoperative pain after 7 days | 7 days after surgery
  Pain intensity was assessed 7 days after surgery using the pain visual analogue scale (VAS) with values ranging from 1 (no pain) to 10 (worst possible pain)
Early postoperative complications | Within 30 days after the surgery
  All complication related to surgery developed within 30 days after the surgery

SECONDARY OUTCOMES:
Chronic Groin pain | After 3 months postoperatively
  Groin pain lasting for more than 3 months after surgery
3 years hernia recurrence rate | within 3 years after surgery
  Unilateral or bilateral - residual or recurrent hernia
Patient's satisfaction score | within 3 years after surgery
  Patient satisfaction was assessed using 1 to 10 scale where: 9-10 means very satisfied, 7-8: satisfied, 6-7: neutral, 4-5: dissatisfied, <4: very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elmessiry, MD, PhD, Principal Investigator — Assistant Professor of Surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarli L, Iusco DR, Sansebastiano G, Costi R. Simultaneous repair of bilateral inguinal hernias: a prospective, randomized study of open, tension-free versus laparoscopic approach. Surg Laparosc Endosc Percutan Tech. 2001 Aug;11(4):262-7. doi: 10.1097/00129689-200108000-00007. PMID 11525372
- [Background] Feliu X, Claveria R, Besora P, Camps J, Fernandez-Sallent E, Vinas X, Abad JM. Bilateral inguinal hernia repair: laparoscopic or open approach? Hernia. 2011 Feb;15(1):15-8. doi: 10.1007/s10029-010-0736-2. Epub 2010 Oct 21. PMID 20960019